CLINICAL TRIAL: NCT01303419
Title: A Multicenter, Open-Label, Crossover Trial to Assess Non-Inferiority of Dual Energy Contrast-Enhanced Digital Mammography (DE-CEDM) Compared to Contrast-Enhanced Breast Magnetic Resonance Imaging (CE-BMRI) for Identifying a Change in Patient Management in Women With Newly Diagnosed Breast Cancer
Brief Title: Contrast-Enhanced Digital Mammography (CEDM) for Identifying a Change in Management of Women With Newly Diagnosed Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor determined there was sufficient material collected to answer the study questions.
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DE-CEDM-001
Record Dates: First submitted 2011-02-18; First posted 2011-02-24 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer
Keywords: mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CE-BMRI (Experimental): Subject will undergo bilateral CE-BMRI as per usual clinical practice within 30 days after the new breast cancer diagnosis. Subject will then undergo bilateral DE-CEDM examination within 8 weeks after the CE-BMRI exam.
  Interventions: Device: CE-BMRI; Device: DE-CEDM

INTERVENTIONS:
Device: CE-BMRI — Contrast-enhanced breast imaging using Magnetic Resonance
Device: DE-CEDM — Breast imaging using Dual-energy, contrast-enhanced digital mammography

SUMMARY:
Enrolled women will undergo a bilateral Contrast-Enhanced Breast Magnetic Resonance Imaging (CE-BMRI) as per usual clinical practice within 30 days of breast cancer diagnosis. Up to 8 weeks after the CE-BMRI exam, subjects will undergo a Dual Energy Contrast Enhanced Digital Mammograph (DE-CEDM).

DETAILED DESCRIPTION:
Enrolled women will undergo a bilateral Contrast-Enhanced Breast Magnetic Resonance Imaging (CE-BMRI) as per usual clinical practice within 30 days of breast cancer diagnosis. Up to 8 weeks after the CE-BMRI exam, subjects will undergo a Dual Energy Contrast Enhanced Digital Mammograph (DE-CEDM). Maximum lesion size was compared between the two imaging types. Subject data from both scans was planned to be included in a multi-reader evaluation; however, due to premature stop of the study, multi-reader data was not collected.

ELIGIBILITY:
Inclusion Criteria:

* Woman 21 years of age or older
* The subject is able and willing to comply with study procedures and signed and dated informed consent is obtained.
* Newly diagnosed with Breast Cancer (DCIS or invasive) identified through core biopsy or fine-needle aspiration (FNA) within last 30 days.
* Will have or have had a bilateral CE-BMRI performed within 30 days AFTER the new breast cancer diagnosis.

Exclusion Criteria:

* Woman who has already had a lumpectomy for the index lesion.
* Woman undergoing neoadjuvant chemotherapy treatment, hormone treatment or radiation therapy.
* Woman who is pregnant or who believe she may be pregnant.
* Woman who has breast implant.
* Woman who has a contraindication to the intravenous use of iodinated or gadolinium-chelated contrast agent (e.g., allergy to either agent or severely impaired renal function).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2010-04; Primary Completion 2012-06-30 (Actual); Study Completion 2012-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Seattle Cancer Care Alliance, Seattle, Washington, United States
- AZ St-Jan Brugge AV, Bruges, Belgium
- Sunnybrook Health Science Centre, Toronto, Canada
- Institut Goustave Roussy, Villejuif, France
- Institut fur Radiologie, Charite, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women 21 years of age or older, with newly diagnosed cancer identified through through core biopsy or fine-needle aspiration (FNA) within the last 30 days and with a bilateral CE-BMRI performed within 30 days of the new breast cancer diagnosis.
Groups:
- CE-BMRI and DE-CEDM Examinations: Subject will undergo bilateral CE-BMRI as per usual clinical practice within 30 days after the new breast cancer diagnosis. Subject will then undergo bilateral DE-CEDM examination within 8 weeks after the CE-BMRI exam.
  CE-BMRI: Contrast-enhanced breast imaging using Magnetic Resonance
  DE-CEDM: Breast imaging using Dual-energy, contrast-enhanced digital mammography
Period: Overall Study
Arm/Group | CE-BMRI and DE-CEDM Examinations
Started | 224 (Subjects who met all Inclusion and none of the Exclusion criteria)
Completed | 128
Not Completed | 96
Not completed — Discontinuation of study | 60
Not completed — Did not complete both imaging methods | 5
Not completed — Did not meet all I/E after screening | 31

BASELINE CHARACTERISTICS:
Population: All participants enrolled in study.
Arm/Group | CE-BMRI and DE-CEDM Examinations
Number analyzed (Participants) | 224
Age, Customized [Count of Participants; unit: Participants]
  Subjects age 21 years or older | 224
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224
  Male | 0
Region of Enrollment [Number; unit: participants]
  Canada | 5
  Belgium | 29
  United States | 13
  France | 59
  Germany | 118

OUTCOME MEASURES:

1. Primary Outcome: Completion of CE-BMRI and DE-CEDM
Description: Subjects have completed both CE-BMRI and DE-CEDM scan types
Time Frame: Approximately 8 weeks
Population: Total number of participants enrolled in the study
Measure: Count of Participants; unit: Participants
Arm/Group | CE-BMRI and DE-CEDM Examinations
Number analyzed (Participants) | 224
Participants
  Subjects completing both scan types | 128
  Subjects did not complete both scan typess | 96

2. Primary Outcome: Average Maximum Lesion Size by CE-BMRI Scan
Description: Average maximum lesion size when scanned using CE-BMRI
Time Frame: Within 1 week of CE-BMRI scan
Population: All subjects who completed both CE-BMRI and DE-CEDM examinations
Measure: Mean (Full Range); unit: millimeters (mm)
Arm/Group | CE-BMRI and DE-CEDM Examinations
Number analyzed (Participants) | 128
millimeters (mm) | 28.8 [6.0 to 110.0]

3. Primary Outcome: Average Maximum Lesion Size by DE-CEDM
Description: Average maximum lesion size when scanned using DE-CEDM
Time Frame: Within 1 week of DE-CEDM scan
Population: All subjects who completed both CE-BMRI and DE-CEDM examinations
Measure: Mean (Full Range); unit: millimeters (mm)
Arm/Group | CE-BMRI and DE-CEDM Examinations
Number analyzed (Participants) | 128
millimeters (mm) | 30.5 [5.0 to 150.0]

4. Primary Outcome: Average Maximum Lesion Size by Histology Outcome
Description: Average maximum lesion size as described in histology report.
Time Frame: Approximately 1 week; upon completion of histology report
Population: Subjects who underwent CE-BMRI and DE-CEDM
Measure: Mean (Full Range); unit: millimeters (mm)
Arm/Group | CE-BMRI and DE-CEDM Examinations
Number analyzed (Participants) | 128
millimeters (mm) | 28.2 [4.0 to 169.0]

5. Primary Outcome: Multi-reader Evaluation of Images
Description: Multi-reader evaluation of images and comparison between CE-BMRI vs. DE-CEDM to determine which technology can more precisely measure cancer size as determined by pathological examination was planned. This was not conducted due to premature stop of the study.
Time Frame: This outcome did not occur due to premature study stop.
Population: Study was prematurely stopped.
Arm/Group | CE-BMRI and DE-CEDM Examinations
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Duration of scan - approximately 1 hour
Arm/Group | CE-BMRI and DE-CEDM Examinations
All-Cause Mortality (participants affected / at risk) | 0/224
Serious Adverse Events (participants affected / at risk) | 0/224
Other Adverse Events (participants affected / at risk) | 9/224
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CE-BMRI and DE-CEDM Examinations (N=224)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
extravasation (General disorders) | 4 (4)
Allergy to contrast media (Immune system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2)
Panic attack (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No